CLINICAL TRIAL: NCT05377320
Title: PAtient Similarity for Decision-Making in Prevention of Cardiovascular Toxicity (PACT): A Feasibility Study
Status: Not yet recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Yee Chung Cheng, Associate Professor, Medical College of Wisconsin
Other Study IDs: PRO00039290
Record Dates: First submitted 2022-04-29; First posted 2022-05-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure; Coronary Artery Disease; Peripheral Artery Disease; Ischemia; Hypertension; Diabetes Mellitus; Cardiomyopathies; Cardiotoxicity
Keywords: clinical decision aid; cancer; cardiac dysfunction; cardio-oncology; artificial intelligence; machine learning; adverse events
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease; Peripheral Arterial Disease; Ischemia; Hypertension; Diabetes Mellitus; Cardiomyopathies; Cardiotoxicity; Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Clinical Decision Aid Group: In this group, physicians will use standard care plus the clinical decision aid.
  Interventions: Other: Clinical Decision Aid
- Control Group: In this group, physicians will use standard care only.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Clinical Decision Aid — The clinical decision aid tool will be used at the subject's first visit (Week 0), Week 12 and Week 24.
  Groups: Clinical Decision Aid Group
Other: Standard Care — Cardiology clinic visits will take place at the subjects first visit (Week 0), Week 12 and Week 24.
  Groups: Control Group

SUMMARY:
This is a single-center, double-arm, open-label, randomized feasibility study that will determine whether a novel clinical decision aid accessed via the electronic health record will be acceptable to both cancer survivors and their cardiologists, will favorably impact appropriate medication use and cardiac imaging surveillance, and will improve clinician and patient decision-making, perception, and behavior towards cardioprotective medication usage and cardiovascular disease imaging utilization.

DETAILED DESCRIPTION:
For this feasibility study, the researchers will create the clinical decision aid and test the central hypothesis that this novel clinical decision aid accessed via the electronic health record will be acceptable to both cancer survivors and their cardiologists and will favorably impact appropriate medication use and cardiac imaging surveillance. The hypothesis is supported by preliminary data suggesting that an initial and rudimentary version of the clinical aid increases appropriate medication use and imaging follow-up in cardio-oncology patients. Success will be determined by ≥85% of clinic visits using the clinical decision aid resulting in pursuit of medication use and cardiac imaging surveillance patterns commensurate with recommendations specific to cancer survivors, with overall rates the same or higher than the group without the clinical decision aid, as well as overall favorable patient and physician focus group comments and survey responses.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years with a history of cancer.
2. Have not previously visited a cardiologist to assess cardiovascular risk after cancer diagnosis.
3. Clinically at intermediate, high, or very high risk for cardiovascular diseases determined based on imprecise clinical risk models, such as those used for cardiac dysfunction.
4. Ability to understand a written informed consent form, and willing to sign it prior to study registration.

Exclusion Criteria:

1. Patient <18 years.
2. Without a personal history of cancer.
3. Existing cardiomyopathy diagnosed after cancer diagnosis.
4. Documented cognitive impairment.
5. Patient or patient representative who is unable and unwilling to sign the informed consent form.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cancer survivors at intermediate, high, or very high risk for developing cardiovascular disease will pursue a cardio-oncology visit.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Medication use | Week 0
  The number of subjects in which medication use pursued is consistent with current medical society recommendations appropriate for the subject.
Medication use | Week 12
  The number of subjects in which medication use pursued is consistent with current medical society recommendations appropriate for the subject.
Medication use | Week 24
  The number of subjects in which medication use pursued is consistent with current medical society recommendations appropriate for the subject.
Imaging surveillance | Week 0
  The number of subjects in which imaging surveillance pursued is consistent with current medical society recommendations appropriate for the subject.
Imaging surveillance | Week 12
  The number of subjects in which imaging surveillance pursued is consistent with current medical society recommendations appropriate for the subject.
Imaging surveillance | Week 24
  The number of subjects in which imaging surveillance pursued is consistent with current medical society recommendations appropriate for the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Yee Chung Cheng, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown SA, Chung BY, Doshi K, Hamid A, Pederson E, Maddula R, Hanna A, Choudhuri I, Sparapani R, Bagheri Mohamadi Pour M, Zhang J, Kothari AN, Collier P, Caraballo P, Noseworthy P, Arruda-Olson A; Cardio-Oncology Artificial Intelligence Informatics and Precision Equity (CAIPE) Research Team Investigators. Patient similarity and other artificial intelligence machine learning algorithms in clinical decision aid for shared decision-making in the Prevention of Cardiovascular Toxicity (PACT): a feasibility trial design. Cardiooncology. 2023 Jan 23;9(1):7. doi: 10.1186/s40959-022-00151-0. PMID 36691060
- [Derived] Brown SA, Fang MZ, Sparapani R, Zhou Y, Osinski K, Taylor B, Yu D, Blessing J, Shah R, Collier P, BagheriMohamadiPour M, Zhang J, Kothari A, Echefu G, Rickards J, Otto C, Sanchez Z, Olson J, Arruda-Olson A, Cheng YC, Cheng F; Cardio-Oncology Artificial Intelligence Informatics and Precision Equity, and Patient Similarity Algorithms in the Prevention of Cardiovascular Toxicity Research Team Investigators. PrevCardioOncAI: Machine Learning Algorithms for Predicting Cardiovascular Disease in Cancer Survivors. J Am Heart Assoc. 2025 Dec 16;14(24):e030363. doi: 10.1161/JAHA.123.030363. Epub 2025 Dec 11. PMID 41378455
- [Derived] Brown SA, Hamid A, Pederson E, Bs AH, Maddula R, Goodman R, Lamberg M, Caraballo P, Noseworthy P, Lukan O, Echefu G, Berman G, Choudhuri I; Cardio-Oncology Artificial Intelligence Informatics & Precision Equity (CAIPE) and Patient Similarity Algorithms in the Prevention of Cardiovascular Toxicity (PACT) Research Team Investigators. Simplified rules-based tool to facilitate the application of up-to-date management recommendations in cardio-oncology. Cardiooncology. 2023 Oct 27;9(1):37. doi: 10.1186/s40959-023-00179-w. PMID 37891699